CLINICAL TRIAL: NCT02561091
Title: Efficacy and Safety of AM-111 in the Treatment of Acute Inner Ear Hearing Loss
Brief Title: AM-111 in the Treatment of Acute Inner Ear Hearing Loss
Acronym: HEALOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Auris Medical AG (Industry)
Responsible Party: Sponsor
Organization: Auris Medical, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AM-111-CL-13-01
Record Dates: First submitted 2015-09-23; First posted 2015-09-25 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Hearing Loss
Keywords: Deafness; Hearing Loss, Sensorineural; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases; Sensation Disorders; Signs and Symptoms; Hearing and Speech impairment; Hearing Loss, Unilateral
MeSH Terms: conditions — Hearing Loss; Deafness; Hearing Loss, Sensorineural; Ear Diseases; Hearing Disorders; Otorhinolaryngologic Diseases; Sensation Disorders; Signs and Symptoms; Speech Disorders; Hearing Loss, Unilateral | interventions — D-JNKI-1

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo gel for intratympanic use
  Interventions: Other: Placebo
- AM-111 0.4 mg/ml (Experimental): AM-111 gel for intratympanic use (0.4 mg/ml AM-111)
  Interventions: Drug: AM-111 0.4 mg/ml
- AM-111 0.8 mg/ml (Experimental): AM-111 gel for intratympanic use (0.8 mg/ml AM-111)
  Interventions: Drug: AM-111 0.8 mg/ml

INTERVENTIONS:
Other: Placebo
  Arms: Placebo
Drug: AM-111 0.4 mg/ml
  Arms: AM-111 0.4 mg/ml
Drug: AM-111 0.8 mg/ml
  Arms: AM-111 0.8 mg/ml

SUMMARY:
The purpose of this research study is to test the effectiveness and safety of the study drug, AM-111. AM-111 is tested for the treatment of sudden sensorineural hearing loss where the cause is unknown.

DETAILED DESCRIPTION:
This phase III study is assessing the drug's safety and is aiming to demonstrate efficacy of intratympanic AM-111 injections in the treatment of severe to profound idiopathic sudden sensorineural hearing loss (ISSNHL). The active pharmaceutical ingredient of AM-111 is the JNK inhibitor (D-JNKI-1), a synthetic peptide consisting of 31 D-amino acids, which acts as a c-Jun N-terminal kinase (JNK) ligand.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral ISSNHL with onset within 72 hours prior to study treatment;
2. Mean hearing threshold of equal to or worse than (≥) 60 dB averaged across the 3 most affected contiguous air conduction audiometric pure tone frequencies ("pure tone average", PTA);*
3. Mean hearing loss of equal to or worse than (≥) 40 dB averaged across the air conducted PTA frequencies compared with the unaffected contralateral ear or reference values from a pre-existing audiogram or ISO 7029;2000 norm values in case of asymmetric hearing prior to the ISSNHL incident;
4. Age ≥ 18 and ≤ 65 years on the day of screening;

Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

1. Bilateral ISSNHL;
2. Acute hearing loss from noise trauma, barotrauma or head trauma;
3. History of autoimmune hearing loss, radiation-induced hearing loss, endolymphatic hydrops or Menière's disease in the affected ear;
4. History of chronic inflammatory or suppurative ear disease or cholesteatoma in the affected ear;
5. History of acoustic neuroma or other retrocochlear damage in the affected ear;
6. History of otosclerosis in the affected ear;
7. Suspected perilymph fistula or membrane rupture in the affected ear;
8. Congenital hearing loss;
9. History of ISSNHL in the past 2 years;
10. Otitis media or otitis externa that is ongoing or ended within 7 days prior to study treatment;

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2015-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Pure tone average (PTA; average of the hearing threshold of three contiguous most affected hearing frequencies in dB) | Day 28
  Assessment with pure tone audiometry/ Measurement at 8 frequencies/ Final outcome is the absolute improvement in PTA from D0 to D28

CONTACTS AND LOCATIONS:
Locations (1):
- Please check link to study webpage below for more study sites, Sofia, Bulgaria

REFERENCES:
- See also: Link to Result entry in clinicaltrialsregister.eu — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-002077-21/results
- See also: Link to peer-reviewed publication of study — https://pubmed.ncbi.nlm.nih.gov/31083077/